CLINICAL TRIAL: NCT06417879
Title: Attitude And Practice of Egyptian Dental Practitioners Regarding Restoration Repair: A Cross-Sectional Study
Brief Title: Attitude And Practice of Egyptian Dental Practitioners Regarding Restoration Repair
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Habiba Hassan Mostafa Hosni, Masters candidate at faculty of dentistry Cairo University, Cairo University
Other Study IDs: 14422021484209
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Practice; Attitude; Dental Restoration Repair
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross-sectional study with an aim to evaluate the variations in self-reporting attitude and practice of restoration repair among Egyptian dental practitioners utilizing a survey questionnaire.

It is undeniable that "Minimally invasive dentistry" nowadays offers solutions to prolong the longevity of resin composite restoration with adhesive technology. Due to the limited lifespan of dental restorations, defects are more prone to occur in the existing restorations and thus require dental treatment. it was stated in the literature that repairing could offer better advantages even though replacement of a restoration is a more common choice by many clinicians.

Since the concept of preserving tooth structure nowadays plays a major part in dental practice, invistigators need to understand where Egyptian dental practitioners stand in understanding and applying the concept of restoration repair. Assessment of knowledge and the missing data regarding the concept of repair that dentists in Egypt have could help understand their awareness in applying conservatism in daily practice. There were some research about knowledge, attitude and practice of restoration repair in of dental practitioners in other countries, but little was known in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian dental practitioners that have completed their bachelor's degree, internship, have practice license and registered in the Egyptian Dental Syndicate.

Exclusion Criteria:

* Undergraduate dental students
* Dental practitioners that are still in internship
* Dental practitioners that don't have their practice license yet.
* Dental practitioners that are not registered in the Egyptian Dental Syndicate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian dental practitioners that have completed their bachelor's degree, internship, have practice license and registered in the Egyptian Dental Syndicate.
Sampling Method: Probability Sample
Enrollment: 316 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Practice of Egyptian dental practitioners toward repair restoration | After data collection (4 months)
  Survey Questionnaire (Percentages)
Attitude of Egyptian dental practitioners toward repair restoration | After data collection (4 months)
  Survey Questionnaire (Percentages)